CLINICAL TRIAL: NCT04608877
Title: Take 5 + Audio Clip Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000027445
Record Dates: First submitted 2020-03-17; First posted 2020-10-29 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Abuse, Child; Crying; Parent-Child Relations
MeSH Terms: conditions — Crying

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Take 5 Only (Placebo Comparator): Parent will only receive the 5 discrete safety steps for infant crying
  Interventions: Behavioral: Take 5 Only
- Take 5 and Audio Clip (Experimental): Parent will receive the 5 discrete safety steps for infant crying and listen to the audio clip of infant crying and public service announcement message
  Interventions: Behavioral: Take 5 and Audio Clip

INTERVENTIONS:
Behavioral: Take 5 and Audio Clip — Parent will receive the 5 discrete safety steps for infant crying and listen to the audio clip of infant crying and public service announcement message
  Arms: Take 5 and Audio Clip
Behavioral: Take 5 Only — Parent will only receive the 5 discrete safety steps for infant crying
  Arms: Take 5 Only

SUMMARY:
At Yale New Haven Hospital, parents on the postpartum ward receive a Take 5 program to help train and prepare parents for strategies to manage their infant's crying. Inconsolable crying is a leading cause for abusive head trauma (AHT) in infants, and the Take 5 program has proven effective in reducing rates of AHT. However, it is also important to examine new ways of improving AHT preventative programs to optimize outcomes for infants. The purpose of this proposal is to determine whether adding a one-minute audio-clip of an infant crying, which specifically addresses AHT, to the Take 5 message given to parents of newborns on the postpartum floor of the hospital strengthens the preventive message. This is a randomized controlled trial (RCT) of parents on the postpartum ward; half will receive just Take 5, and the other half will receive the audio-clip and Take 5. Our hypotheses to be tested are that relative to parents who had Take 5 alone, those parents who hear the audio-clip before learning Take 5 will:

1. Have higher HR/BPs and higher negative affect after the training session
2. Be more likely to remember use Take 5 when they became frustrated with their infant's crying when followed up 6 weeks later.
3. Be more likely to tell other people about Take 5 and be more likely to say Take 5 was useful.

DETAILED DESCRIPTION:
The purpose of this proposal is to determine whether adding the one-minute audio-clip of an infant crying to the Take 5 message given to parents of newborns on the postpartum floor of the hospital strengthens the preventive message. To do this, a randomized controlled trial (RCT) will be conducted. The investigators would like to determine if the anticipatory guidance of Take 5 is strengthened by hearing a 1-minute audio-clip of an infant crying followed by a preventive message about abusive head trauma, which was used as a radio public service announcement in Milwaukee, Wisconsin as part of a non-programmatic effort to reduce the rates of AHT and is used with permission. All families in the post-partum unit are eligible to have the Take 5 message as part of their anticipatory guidance before newborn hospital discharge.

Randomization will be done based on the postpartum day of life. If the infant's postpartum date of life is an even number, parents will get Take 5 only; for odd numbers, they would get Take 5 and the audio PSA.

For both groups, three baseline self-report measures will be obtained: the Reflective Functioning Questionnaire, the Parenting Stress Index, and the Emotion Regulation Questionnaire; and 5 measures will be obtained at baseline and after the recording: blood pressure, heart rate, and affect descriptors. Affective descriptors include the Positive and Negative Affective Scale and Likert-scales of self-reported levels of stress and frustration.

After the baseline measures have been obtained, all parents will receive the current standard of care -- Take 5, the safety plan for crying. For infants born on odd days, the audio recording will be played before the parent is taught Take 5. For infants born on even days, the parent will receive Take 5. After obtaining the post-recording self-report and physiological measures, we will also ask parents using a 5-point Likert the extent to which Take 5 (both conditions), and the audio recording (odd condition only) might impact them and the caregiving practices related to their infant. About six weeks after, each parent will be contacted by phone and asked about his/her memory of the recording, how many and whom they told about the recording, and what effect if any the recording had on their self-awareness about crying and about their behaviors toward their infant. We will use a 5-point Likert scale to have parents who heard the audiotape before being taught. Take 5 describe the extent to which the recording had impacted them and their infant caregiving practices. We will also ask all parents what impact Take 5 had on their caregiving using 5-point Likert scales as well. The research protocol in the hospital should take no longer than 25 minutes. This second (telephone) interview will also be audio recorded, and then a transcript will be made for analysis. A scripted questionnaire will be used to conduct a telephone interview (see attached Interview.docx). This second interview should last approximately 10 minutes.

Demographic data to be collected on the sample includes parental age, parental sex, parental ethnicity, marital status, the highest level of education (in years), number of children, age of the youngest child, age of other children (if any), number of people living in the household. We will also collect two contact phone numbers and an email address for the participant. We will also collect information on child outcomes, namely: mode of delivery, gestational age, gestational birth weight, and any complications following delivery.

ELIGIBILITY:
Inclusion Criteria:

- parent of singleton newborn on the postpartum floor of the YNHH

Exclusion Criteria:

* presence of severe psychiatric or substance-related symptoms requiring in-patient psychiatric hospitalization or ambulatory detoxification
* persons incapable of giving informed consent
* insufficient English fluency
* maternal medical complication from delivery (e.g eclampsia, postpartum hemorrhage or infection)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Usage of Take 5 | 1 year
  Participants will be asked if they used Take 5

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Bechtel, MD, Principal Investigator — Professor of Pediatrics (Emergency Medicine) and of Emergency Medicine
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: August 2023